CLINICAL TRIAL: NCT03685253
Title: Nicotinamide Riboside in Diabetic Polyneuropathy
Brief Title: Nicotinamide Riboside for Diabetic Neuropathy
Acronym: NiRiD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Completed the pilot study and grant funding not obtained to continue to the main phase 2 study. The pilot study did not show a statistical significance in the primary or secondary outcome measures.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, James W. Russell, MD, MS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00080331
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Neuropathy Peripheral
Keywords: diabetes; neuropathy; treatment; drug
MeSH Terms: conditions — Diabetes Mellitus | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants randomized to placebo will take 2 capsules by mouth twice a day for 6 months. The placebo capsules are matched to the NR capsules.
  Interventions: Drug: Placebo
- Niagen® (Experimental): Participants randomized to Niagen® (3-(Aminocarbonyl)-1-β-D-ribofuranosyl-pyridinium chloride - NR) will take 250 mg capsules. Participants will take 2 capsules by mouth twice a day (1000 mg) for 6 months
  Interventions: Drug: Niagen

INTERVENTIONS:
Drug: Niagen — Niagen® (3-(Aminocarbonyl)-1-β-D-ribofuranosyl-pyridinium chloride - NR) will be the experimental treatment, at a dose of 1000 mg/day taken as two 250 mg capsules twice daily for 6 months.
  Other Names: Nicotinamide Riboside; 3-(Aminocarbonyl)-1-β-D-ribofuranosyl-pyridinium chloride
  Arms: Niagen®
Drug: Placebo — Placebo capsules matched to the experimental drug and taken orally as 2 capsules twice daily for 6 months.
  Arms: Placebo

SUMMARY:
At the current time there is no effective disease modifying therapy for diabetic neuropathy (DN). The proposed study design employs a quantifiable early measure of DN, intraepidermal nerve fiber density (IENFD), allowing for accurate assessment of actual nerve fiber density. Preclinical data supports the use of Niagen® (3-(Aminocarbonyl)-1-β-D-ribofuranosyl-pyridinium chloride - NR) as a potential therapy for diabetic neuropathy. Phase I data indicates safety in humans. This study seeks to investigate the use of Niagen® (NR) as a potential treatment for diabetic neuropathy in subjects with type 2 diabetes mellitus or impaired glucose tolerance over a 6 month period. The endpoint measures in addition to the IENFD with determine changes in clinical and electrophysiological outcomes, quality of life and biochemical measures.

DETAILED DESCRIPTION:
At the current time there is no effective disease modifying therapy for diabetic neuropathy (DN). Previous failed trials of therapy have often targeted individuals with advanced, severe neuropathy. There is a particularly strong incentive to treat neuropathy early in its course while the severity is still mild and to target participants who have impaired glucose tolerance (IGT) or who have well controlled type 2 diabetes mellitus (T2DM). The proposed study design employs a quantifiable early measure of DN, intraepidermal nerve fiber density (IENFD) of the thigh, allowing for accurate assessment of actual nerve fiber density over time, while also incorporating measures of pain and quality of life. Preclinical data supports the use of NR as a potential therapy for diabetic neuropathy. Phase I data indicates safety in humans.

The most common form of diabetes mellitus, T2DM, is projected to affect an estimated 366 million people worldwide by 2030. The lifetime incidence of polyneuropathy is approximately 45% and neuropathy of any type approximately 59% of in patients with T2DM. Studies of nerve conduction tests performed at the time of diabetes mellitus diagnosis demonstrate that neuropathy is already present in patients when the neuropathy is still subclinical. Furthermore, DN leads to severe morbidity, high mortality, major physical disability, poor quality of life, and high cost with estimated total annual costs of $22 billion (www.diabetes.org). Due to the complex structure and anatomy of the peripheral nervous system, DN presents with a very broad spectrum of clinical symptoms and deficits, including severe pain, sensory deficits, foot ulcers and amputations. Despite the high morbidity associated with DN, most randomized clinical trials evaluating therapies for established DN have been disappointing. To date there is no pathogenetic treatment for this condition. Currently, tight glycemic control is the only convincing strategy to prevent or delay the development of DN in patients with type 1 diabetes mellitus. There is less convincing evidence that tight glycemic control improves neuropathy with T2DM.

DN is a diffuse, symmetrical injury to the entire peripheral nervous system. The smallest Aδ thinly-myelinated fibers and the unmyelinated C-fibers are likely the earliest to undergo damage in the natural history of DN. These fibers mediate pain, temperature discrimination, touch perception and autonomic responses, and constitute over 80% of peripheral nerve fibers. When determining the effect of a therapeutic intervention in DN it is important to utilize outcome measures that best identify change in disease. Although both large and small fiber neuropathy occur in T2DM, a small-fiber neuropathy is more common. Importantly, developing appropriate endpoints has been a problem in DN because many of the endpoints have proved too insensitive in clinical trials. For example, there is a need to establish content validity in clinical scales. IENFD is a sensitive and reliable measure in determining change in early DN. Furthermore, IENFD directly correlates with increasing DN severity, and is safe as easy to perform and IENFD currently represents a gold standard in measuring change in small fiber neuropathy. Thus, IENFD was selected as the most appropriate endpoint measure in this clinical trial. The morphometric quantification of IENFD is easily measured from a skin biopsy and this is used as part of routine clinical practice. The skin biopsy is a minimally invasive procedure and less than 1% of participants have mild adverse events such as bleeding, infection, or delayed healing. Inter-observer variability for the assessment of IENFD demonstrates good agreement, especially with assessment at the thigh. Patient refusal rate for this procedure is minimal (less than 1 %).

This is a phase II, single center, randomized, double-blind, placebo-controlled clinical trial to evaluate the effect of NR compared to placebo on measures of small fiber neuropathy in participants with IGT or T2DM and mild DN. Participants with be randomly assigned to either NR 0.5 grams twice a day (total 1 gram/day) or matched placebo in a 1:1 ratio. Participants in the active group will start with a 1 gram/day dose because of the very low risk of adverse events with NR. The 1 gram/day dose will be taken continuously for 6 months. In addition (if they have not already received this information) all participants will be given general diabetic nutritional advice and general advice to exercise for approximately 150 minutes per week. This represents current standard of care information provided to all patients with impaired glucose regulation and DN.

Primary efficacy measure: change in the thigh IENFD at 6 months compared to baseline. Secondary efficacy measure: change in the distal leg IENFD at 6 months compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Impaired glucose tolerance or controlled type 2 diabetes mellitus at the time of screening or within three months of screening*.
2. The hemoglobin A1c may be normal, but should be less than 9%.
3. If diabetic participants are on medication, they should be stable on medication for at least 3 months prior to entering the study. Addition or change in antidiabetic medication (if on medication) after enrollment does not affect participation or group assignment.
4. Impaired glucose regulation is the most likely cause of the neuropathy.
5. Mild diabetic polyneuropathy as defined by the Toronto Diabetic Neuropathy Expert Group consensus criteria.
6. Age 30 (to exclude patients with type 1 diabetes) to 80 years inclusive.
7. Medically stable at the time of enrollment.
8. Willing to accept randomization assignment and compliance with the study procedures.

Exclusion Criteria:

1. Women of childbearing potential must be using an acceptable method of contraception to prevent pregnancy when they are enrolled in the study.
2. Patient must agree to take an alternative medication to Warfarin or Factor X inhibitors when undergoing a skin biopsy.
3. Neuropathy due to factors other than type 2 diabetes mellitus based on careful clinical and laboratory evaluation by the study physicians.
4. Abnormal liver function tests, including alanine transaminase, aspartate transaminase, alkaline phosphatase, and bilirubin.
5. Current severe medical conditions that are active on the day of screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Thigh Intraepidermal Nerve Fiber Density | 6 months.
  Change in the proximal thigh Intra-Epidermal Nerve Fiber Density as assessed by skin biopsy. Smaller values indicate worse neuropathy. Normative ranges depend on age and gender.

SECONDARY OUTCOMES:
Distal lower limb intraepidermal nerve fiber density | 6 months.
  Change in the distal leg Intra-epidermal Nerve Fiber Density as assessed by biopsy. Smaller values indicate worse neuropathy. Normative ranges depend on age and gender.

OTHER OUTCOMES:
Modified Toronto Clinical Neuropathy Scale | 6 months.
  Modified Toronto Clinical Neuropathy Scale to assess clinical symptoms and signs of diabetic neuropathy
Total Neuropathy Score (Clinical) | 6 months.
  Total Neuropathy Score (Clinical)
The Neuropathy Total Symptom Score (NTSS-6) | 6 months.
  The Neuropathy Total Symptom Score ranges from 0 to 21.96 points with higher scores indicating a worse symptom score
Pain Quality Assessment Scale | 6 months.
  To evaluate the neuropathic pain and non-neuropathic pain. The Pain Quality Assessment Scale was developed from the neuropathy Pain Scale and is a 20 item scale that assesses both neuropathic pain and non-neuropathic pain. Higher score indicate worse pain.
Survey of Autonomic Symptoms | 6 months.
  Survey of Autonomic Symptoms to assess symptoms of peripheral autonomic function. The scale varies depending on gender. Higher scores indicate higher levels of autonomic symptoms.
Neuro Quality of Life Measure | 6 months.
  This measures quality of life and is an 11 item scale with each item scored from 0 to create an aggregate scale. High scores are worse.
Nerve Conduction Studies | 6 months.
  Nerve Conduction Studies to assess changes in nerve conduction. The amplitudes of the sural sensory, fibular motor, tibial motor and their respective distal latencies, and conduction velocities are obtained. Data will be used from individual measurements and using a mega score of combined variables. Lower scores may indicate neuropathy.
Cardiac Autonomic Neuropathy | 6 months.
  The expiration:inspiration ratio will be measured. Normative data varies depending on age, gender and other factors. Lower scores may indicate cardiac autonomic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: James W Russell, MD, Principal Investigator — University of Maryland School of Medicine & Department of Veterans' Affairs
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No